CLINICAL TRIAL: NCT06527378
Title: The Role and Applications of Artificial Intelligence in Dental Implant Planning
Brief Title: Artificial Intelligence in Dental Implant Planning
Acronym: AIDENT
Status: Completed | Type: Observational
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, Principal Investigator, University of Bari Aldo Moro
Other Study IDs: AI in Dentistry
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Edentulous Alveolar Ridge; Edentulous Mouth; Tooth Loss
Keywords: Artificial Intelligence in Implantology; AI in Dental Implantology; Machine Learning in Dental Implantology; Deep Learning in Implant Dentistry; Robotics in Dental Implantology; AI-Based Implant Planning
MeSH Terms: conditions — Mouth, Edentulous; Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: AI in implant planning — Assessment of Current Technology for Supporting Implant Planning

SUMMARY:
Artificial intelligence (AI) is revolutionizing the dentistry, offering new opportunities to improve the precision and efficiency of implantology. This study aims to evaluate the current evidence on the use of AI in implant planning assessment

DETAILED DESCRIPTION:
The analysis was conducted through electronic search engines, using a combination of relevant keywords, including "artificial intelligence implantology," "AI implant planning," "AI dental implant," and "implantology artificial intelligence." Selected articles will carefully re-viewed to identify studies reporting data on the effectiveness of AI in implant planning.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent 3D or 2D radiological examinations for implant-prosthetic rehabilitation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with edentulous ridges who need fixed prosthetic rehabilitation
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Valuation on the diagnosis of anatomical structures | 1 month
  The primary focus is on evaluating the AI tools to evalue the quality and dimensions of the bone and ensuring the safe placement of implants by identifying and preserving critical structures such as nerves and the max-illary sinus.

CONTACTS AND LOCATIONS:
Locations (1):
- Giuseppe D'Albis, Mola di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macri M, D'Albis V, D'Albis G, Forte M, Capodiferro S, Favia G, Alrashadah AO, Garcia VD, Festa F. The Role and Applications of Artificial Intelligence in Dental Implant Planning: A Systematic Review. Bioengineering (Basel). 2024 Jul 31;11(8):778. doi: 10.3390/bioengineering11080778. PMID 39199736